CLINICAL TRIAL: NCT00523510
Title: Feasibility and Pilot Efficacy of Flash-heated Breast Milk for Reduction of Maternal-to-Child Transmission of HIV in Tanzania
Brief Title: Feasibility and Pilot Efficacy of Flash-heated Breast Milk to Reduce Maternal-to-Child-Transmission of HIV in Tanzania
Acronym: Flash-heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Thrasher Research Fund (Other); University Research Co, LLC (Industry); California Department of Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200513446; N/A yet
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections
Keywords: breastmilk; perinatal HIV; infant feeding; flash heat; pasteurization; pmtct; HIV; HIV Seronegativity; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feasibility Study (Experimental): HIV positive women [and a smaller number of HIV negative/unknown status (1 for every 3 infected women)] to avoid stigmatizing home-based counseling will be recruited at 1-2 postpartum and provided enhanced home-based infant feeding counseling by community health workers to exclusively breastfeed for 6 months. Mothers will also be told about the option to Flash-heat breastmilk during and after the transition from exclusive breastfeeding. Mothers who choose to Flash-heat will be provided continued home-based counseling and support. Feasibility data will be collected during the time mothers Flash-heat.
  Interventions: Procedure: Infant feeding counseling that includes Flash-heat
- Pilot efficacy (Experimental): We will collect infant health data to monitor and compare health outcomes among 3 groups of infants who had exclusive breast feeding (EBF) for the first months and then either: 1) fed Flash-heated breast milk and complementary foods (n=30), or 2) weaned to replacement foods and NO breast milk (n=15; per standard WHO recommendation for rapid cessation), or 3) continued feeding at the breast and providing other foods and/or fluids, i.e. mixed feeds (n=15; per WHO consensus that breastfeeding continue if replacement feeding is not AFASS94). We will collect infant growth and morbidity data. Infant health outcomes will be compared for the 3 groups noted above. These data will be collected primarily to pilot an efficacy trial.
  Interventions: Procedure: Infant feeding counseling that includes Flash-heat

INTERVENTIONS:
Procedure: Infant feeding counseling that includes Flash-heat — Intensive infant feeding counseling which includes description and demonstration of the WHO recommended option for HIV-infected mothers to pasteurize their breastmilk. Flash-heat pasteurization will be described and demonstrated to interested mothers. More intensive counseling and support will be provided home visits.

SUMMARY:
This study will investigate the feasibility of HIV positive mothers in Tanzania to correctly use the Flash-heat method to pasteurize their breast milk and for how long they are able to do so. The patients will be followed in this study for up to 3 months of Flash-heating their milk. Flash-heated breast milk could be a potential method to reduce mother-to-child transmission of HIV. The investigators will also collect infant health data to pilot a future efficacy trial. The investigators hypothesize that with enhanced home-based infant feeding counseling, mothers will be capable of Flash-heating their breast milk.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends human immunodeficiency virus (HIV) positive mothers in developing countries exclusively breastfeed for the first months of the infant's life followed by early cessation, unless breast milk substitutes are acceptable, feasible, affordable, sustainable, and safe. The weaning period is high risk for such infants due to lack of adequate replacement feeds resulting in malnutrition, growth faltering and susceptibility to diarrheal and respiratory illness from loss of breast milk's immune protection and introduction of contaminated foods and water. In addition, risk of HIV transmission is increased if a mother breastfeeds during weaning due to higher breast milk viral load during this time. Appropriate infant feeding alternatives during and after the high-risk weaning period are urgently needed.

Although heat-treating breast milk is listed by WHO as one method of modifying breast milk, it has not been fully explored. Our preliminary data demonstrate that Flash-heat, a low-technologic home pasteurization method, is capable of inactivating HIV in infected breast milk while maintaining most vitamins and immunoglobulins. This suggests Flash-heating breast milk could be a potential infant feeding option during and after weaning to decrease risk of infant illness and malnutrition.

Clinical staffing shortages in much of Africa, however, limit the ability of doctors, nurses and counselors to provide comprehensive infant feeding counseling to each mother. In light of this, our study will investigate the use of enhanced peer-based infant feeding counseling as a practical approach to improving exclusive breastfeeding durations while we are investigating the feasibility of Flash-heating breast milk. We will collaborate with the US and Tanzania offices of the University Research Co, LLC (URC), who are at the forefront of implementing appropriate infant feeding counseling methods in Africa. We will work with URC, local investigators, and Anna Coutsoudis, who's Safer Breastfeeding Programme in South Africa is considered a model, to provide community health workers with comprehensive infant feeding counseling training. HIV positive mothers (and a small number of HIV negative/status unknown mothers to avoid stigmatizing home-based counseling) who are breastfeeding will be recruited at 1-2 months postpartum at hospitals in Tanzania and provided enhanced counseling to exclusively breastfeed. Trained community health workers will make weekly home visits to support the mothers and collect infant feeding and breast pathology data. When the HIV positive mothers anticipate introduction of complementary foods, the Flash-heat method will be further discussed as an option for during and after transition. Mothers who choose to Flash-heat will be provided home-based support by community health workers and followed for up to 3 months from the time they stop breastfeeding.

This feasibility and pilot efficacy study of Flash-heating breast milk will be used to guide a full-scale efficacy trial in the near future. Specific aims include to: 1) Determine the impact of enhanced home-based training on infant feeding outcomes. Given clinical staffing shortages in Tanzania, the use of community health workers could provide support needed to exclusively breastfeed longer. Rates of initiation and duration of exclusive breastfeeding will be measured. These findings are important to explore effective methods of thoroughly educating the mothers about the risks and benefits of the various infant-feeding alternatives while not increasing the burden facing under-staffed health care workers. 2) Determine uptake of the Flash-heat method and protocol adherence by mothers in their homes. With enhanced support from community health workers, mothers may be able to correctly Flash-heat their milk, suggesting it could be a practical infant feeding method. Uptake of heat treatment and the duration of successful heat treatment will be measured. We will also interview mothers who opt to attempt the method to qualitatively assess the challenges mothers may face in a field setting. 3) Determine safety of Flash-heated breast milk in a field setting. Breast milk samples will be collected and assayed for HIV inactivation and bacterial counts to ensure method safety in field settings. 4) To pilot an efficacy trial of Flash-heat to improve infant health outcomes. Research personnel will monitor infant feeding, growth and morbidity during home visits twice monthly. If infants who receive heat-treated breast milk experience less morbidity and mortality than those fed complementary foods while continuing to breastfeed and those completely weaned to replacement foods, counselors in the future will be better able to inform mothers of risks and benefits of different feeding options.

If this proposed study finds that HIV positive mothers can successfully heat-treat their breast milk, it could be viewed as an HIV-free, safe, nutritious, affordable and available complementary food during and after the weaning phase after EBF.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18, with permanent local residence
* 1-2 months post-partum
* Breastfeeding
* HIV-negative or unknown in 1:3 ratio with HIV-positive
* If HIV positive: having CD4+ > 200, not currently on Antiretroviral Therapy (ART)

Exclusion Criteria:

* Males, females under the age of 18
* Women not 1-2 most postpartum
* Women not breastfeeding
* Women with HIV and CD4+ < 200 OR on Antiretroviral Therapy (ART); And
* Women without permanent local residence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the impact of enhanced home-based training on infant feeding outcomes. | 1 year
To determine uptake (initiation and duration) of the Flash-heat method and protocol adherence by mothers in their homes. | 1 year
To determine the safety of Flash-heated breast milk in a field setting. | 1 year

SECONDARY OUTCOMES:
To pilot an efficacy trial of Flash-heat to improve infant health outcomes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Caroline J Chantry, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Israel-Ballard K, Chantry C, Dewey K, Lonnerdal B, Sheppard H, Donovan R, Carlson J, Sage A, Abrams B. Viral, nutritional, and bacterial safety of flash-heated and pretoria-pasteurized breast milk to prevent mother-to-child transmission of HIV in resource-poor countries: a pilot study. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):175-81. doi: 10.1097/01.qai.0000178929.15904.95. PMID 16186735
- [Background] Israel-Ballard KA, Maternowska MC, Abrams BF, Morrison P, Chitibura L, Chipato T, Chirenje ZM, Padian NS, Chantry CJ. Acceptability of heat treating breast milk to prevent mother-to-child transmission of human immunodeficiency virus in Zimbabwe: a qualitative study. J Hum Lact. 2006 Feb;22(1):48-60. doi: 10.1177/0890334405283621. PMID 16467287
- [Background] Israel-Ballard K, Coutsoudis A, Chantry CJ, Sturm AW, Karim F, Sibeko L, Abrams B. Bacterial safety of flash-heated and unheated expressed breastmilk during storage. J Trop Pediatr. 2006 Dec;52(6):399-405. doi: 10.1093/tropej/fml043. Epub 2006 Sep 27. PMID 17005732
- [Background] Chantry CJ, Abrams BF, Donovan RM, Israel-Ballard KA, Sheppard HW. Breast milk pasteurization: appropriate assays to detect HIV inactivation. Infect Dis Obstet Gynecol. 2006;2006:95938. doi: 10.1155/IDOG/2006/95938. No abstract available. PMID 17093357
- [Background] Israel-Ballard K, Donovan R, Chantry C, Coutsoudis A, Sheppard H, Sibeko L, Abrams B. Flash-heat inactivation of HIV-1 in human milk: a potential method to reduce postnatal transmission in developing countries. J Acquir Immune Defic Syndr. 2007 Jul 1;45(3):318-23. doi: 10.1097/QAI.0b013e318074eeca. PMID 17514015
- [Background] Israel-Ballard KA, Abrams BF, Coutsoudis A, Sibeko LN, Cheryk LA, Chantry CJ. Vitamin content of breast milk from HIV-1-infected mothers before and after flash-heat treatment. J Acquir Immune Defic Syndr. 2008 Aug 1;48(4):444-9. doi: 10.1097/QAI.0b013e31817beb8d. PMID 18614920